CLINICAL TRIAL: NCT04631159
Title: Effectiveness of Health Management of Glycemic Control and Physical Activity in Type 2 Diabetes Mellitus Using Smartphone Application:a Randomized Controlled Trial
Brief Title: Effectiveness of Health Management of Glycemic Control and Physical Activity in Type 2 Diabetes Mellitus Using Smartphone Application
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mei-fang Huang (Other)
Responsible Party: Sponsor-Investigator, Mei-fang Huang, ChangGungMH Certified Diabetes Educator, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202000635B0
Record Dates: First submitted 2020-11-03; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: To Investigate the Effectiveness of Health Management of Glycemic Control and Physical Activity in Type 2 Diabetes Mellitus Using Smartphone Application

STUDY DESIGN:
Intervention Model Description: This study will be a randomized controlled trial. Seventy adults (aged 20 to 60 years) diagnosed with T2DM by the physician will recruited and randomly assigned to the mobile app group and the control group. Both groups will receive education by health professionals at Southern Medical Center and they are required to wear fitness watches to record steps. Mobile app group: patients will need to download and use the Health2Sync app and report blood glucose data weekly, and be monitored and advised by medical personnel. Control group: Patients will be asked to self-manage and there is no intervention during the tracking process. Each subject will be required to measure body composition, blood pressure, blood biochemical analysis (HbA1C, fasting blood glucose, total cholesterol, low-density cholesterol, high-density cholesterol, triglycerides), and number of steps before and after 12 weeks
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile app group (Experimental): They are required to wear fitness watches to record steps ,patients will need to download and use the Health2Sync app and report blood glucose data weekly, and be monitored and advised by medical personnel.
  Interventions: Behavioral: Health2Sync app and report blood glucose data weekly
- Control group (Placebo Comparator): they are required to wear fitness watches to record steps ,patients will be asked to self-manage and there is no intervention during the tracking process.
  Interventions: Other: self-manage

INTERVENTIONS:
Behavioral: Health2Sync app and report blood glucose data weekly — Patients will need to download and use the Health2Sync app and report blood glucose data weekly
  Arms: Mobile app group
Other: self-manage — Patients will be asked to self-manage and there is no intervention during the tracking process
  Arms: Control group

SUMMARY:
Medical cost in Taiwan for management of diabetes has accounted for the top three. Diabetic patients often have poor self-health managements, there by leading to occurrence of complications. investigators team has previously published that medical staff directly instructed to the elderly with diabetes comorbid with knee osteoarthritis by performing elastic band resistance exercise, participants can improve functional activity after 12 weeks of intervention. However, there was a decrease in glycated hemoglobin (HbA1c), but it did not reach a significant improvement.Investigators also found that how to improve the glycemic control, particularly in during the follow-up periods, and how to increase the amount of physical activity of diabetic patients that may affect the changes in glycated hemoglobin. With the rapid development of up-to-date medical technology, medical applications (apps) has emerging developing to aid self-health management by themselves. Therefore, this project will continue to explore the effectiveness of using simple tracking, monitoring, and immediate feedback on the health management of diabetic patients. Although various apps have been adopted for the monitoring of diabetic patients, few medical professionals regularly use smartphone apps to directly supervise diabetic patients to make immediate remote medical intervention regarding blood glucose, medications, blood pressure, body composition, and even monitor physical activity concurrently.

DETAILED DESCRIPTION:
Purpose: To investigate the effectiveness of health management of glycemic control and physical activity in type 2 diabetes mellitus (T2DM) using Smartphone application.

Hypothesis: Clinical medical personnel can monitor data through the mobile app platform and provide personalized lifestyle adjustments based on the information provided by patients, thereby improving patient compliance and effectively self-health management in patients with T2DM. At the same time, through this system, medical personnel can understand the amount of physical activity of the patient during this period, and investigators can promptly encourage patients to reach the set goal of physical activity, which can improve the patient's physical status, so this study can bring a positive effect in both blood glucose and related biomarkers.

Methods: This study will be a randomized controlled trial. Seventy adults (aged 20 to 60 years) diagnosed with T2DM by the physician will recruited and randomly assigned to the mobile app group and the control group. Both groups will receive education by health professionals at Southern Medical Center and participants are required to wear fitness watches to record steps. Mobile app group: patients will need to download and use the Health2Sync app and report blood glucose data weekly, and be monitored and advised by medical personnel. Control group: Patients will be asked to self-manage and there is no intervention during the tracking process.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type2 diabetes
* Age 20 to 60 years old

Exclusion Criteria:

* No smartphone, cannot operation of smartphone
* Unable to move
* Use insulin pump
* Pregnant women
* Diagnosis neuropathy
* Diagnosis retinopathy
* Diagnosis diabetic foot
* Diagnosis severe nephropathy ,
* Diagnosis severe liver disease Cognitive impairment

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline HbA1c through a mobile app. | Change from baseline HbA1c at 3 months

SECONDARY OUTCOMES:
The number of participants who have related every day steps as assessed by Mi Smart Band 4. | Change from baseline at 3 months
  The number of participants who have related per day steps as assessed by Mi Smart Band 4. Achieve the goal value of 7500 steps per day.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Nai-Jen, Study Director — Kaohsiung Medical University Department of Sports Medicine professor
Locations (1):
- Mei-fang Huang, Kaohsiung City, No. 20, Ln. 125, Wenbin Rd., Fengshan Dist.,, Taiwan

IPD SHARING:
Plan to Share IPD: No
Currently in the submission stage ,and then share with other researchers after publication